CLINICAL TRIAL: NCT00948688
Title: Phase 1/2 Study of Vorinostat in Combination With Radiation Therapy and Infusional 5-FU in Patients With Locally Advanced Adenocarcinoma of the Pancreas
Brief Title: Vorinostat With XRT and 5-FU for Locally Advanced Adenocarcinoma of the Pancreas
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Funding was withdrawn after only 10 participants were enrolled
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Brigham and Women's Hospital (Other); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Lawrence S. Blaszkowsky, MD, Assistant Physician, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-114
Record Dates: First submitted 2009-07-27; First posted 2009-07-29 (Estimated); Results first posted 2017-05-10 (Actual); Last update posted 2017-05-10 (Actual); Status verified 2017-03

CONDITIONS: Pancreatic Cancer; Adenocarcinoma of the Pancreas
Keywords: Zolinza
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Radiotherapy; Fluorouracil; Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vorinostat, 5-FU, Radiation Therapy (Experimental): Vorinostat at varying doses; orally, days 1-7, weeks 1-6 5-FU 225 mg/m2/day; intravenous; days 1-5, weeks 1-6 until completion of radiation therapy; Radiation therapy; 180cGy daily Monday-Friday; 28 days of treatment (6 weeks)
  Interventions: Radiation: Radiation therapy; Drug: 5-FU; Drug: Vorinostat

INTERVENTIONS:
Radiation: Radiation therapy — Once per day, 5 days a week for 6 weeks
Drug: 5-FU — Intravenously over 24 hours, 7 days per week during each week of radiation therapy
  Other Names: Efudex, Carac, Fluoroplex, Adrucil
Drug: Vorinostat — Taken orally. Dose will depend upon time of enrollment and how well previous participants tolerated the drug
  Other Names: Zolinza

SUMMARY:
The durg vorinostat (Zolinza) is a type of drug called an histone deacetylase (HDAC) inhibitor. It inhibits a group of enzymes called histone deacetylases. These enzymes help cancer cells survive. By inhibiting these enzymes, vorinostat helps kill cancer cells. In this research study vorinostat will be given along with radiation therapy and the drug 5-FU. This is the first research study in which vorinostat will be given along with radiation therapy and 5-FU. The purpose of this research study is to find the highest dose of vorinostat that can be given safely along with radiation therapy and 5-FU. The investigators will also begin to get information about whether vorinostat combined with radiation and 5-FU may help to treat pancreatic cancer.

DETAILED DESCRIPTION:
* Since we are looking for the highest dose of vorinostat that can be administered safely without severe or unmanageable side effects, not everyone who participates will receive the same dose. The dose will depend upon the number of participants enrolled on the study and how well they have tolerated their doses.
* 5-FU will be given intravenously over 24 hours 7 days per week during each week of radiation therapy. In order for participants to be able to receive the 5-FU as an outpatient, they will need to have central line catheter placed.
* Radiation therapy will be given once per day, 5 days per week, for 6 weeks.
* Vorinostat is taken orally.
* Participants will be seen once per week during the 6 weeks that they are receiving 5-FU, radiation therapy and vorinostat.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven adenocarcinoma of the pancreas
* Evaluable disease
* Must have received 3-4 months of gemcitabine-based chemotherapy and have had stable disease by RECIST criteria. Regimens include:

  * gemcitabine alone
  * gemcitabine and erlotinib
  * gemcitabine and oxaliplatin
  * gemcitabine and cisplatin
  * gemcitabine and capecitabine
* 18 years of age or older
* Life expectancy of greater than 4 months
* ECOG Performance Status 0-1
* Normal organ and marrow function as outlined in the protocol
* Ability to drink at least 2 liters of fluid daily
* Women of child-bearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation
* Patients must be able to swallow capsules

Exclusion Criteria:

* Chemotherapy within 3 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Participants may not be receiving any other study agents
* Known distant metastases to any organ
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to vorinostat or 5-FU
* Patients taking warfarin due to potential interactions of both 5-FU and vorinostat. Low molecular weight heparin should be substituted when appropriate
* Patients who have received upper abdominal radiation therapy which fields would overlap with that determined necessary to treat the primary tumor.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or breastfeeding women
* Individuals with history of a different malignancy are ineligible unless they are deemed by the investigator to be at low risk of recurrence of that malignancy. Patients may not have a concurrent second malignancy.
* Active HIV or hepatitis
* Prior exposure to HDAC inhibitor (except valproic acid, provided there is a 30 day washout period)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-08; Primary Completion 2012-06 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Blaszkowsky, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Vorinostat 200 mg: Vorinostat 200 mg; orally, days 1-7, weeks 1-6 5-FU 225 mg/m2/day; intravenous over 24 hours; days 1-5, weeks 1-6 until completion of radiation therapy; Radiation therapy; 180cGy daily Monday-Friday; 28 days of treatment (6 weeks)
- Vorinostat 100 mg: Vorinostat 100 mg; orally, days 1-7, weeks 1-6 5-FU 225 mg/m2/day; intravenous over 24 hours; days 1-5, weeks 1-6 until completion of radiation therapy; Radiation therapy; 180cGy daily Monday-Friday; 28 days of treatment (6 weeks)
Period: Period 1: 200 mg Vorinostat
Arm/Group | Vorinostat 200 mg | Vorinostat 100 mg
Started | 4 | 0
Completed | 2 | 0
Not Completed | 2 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Protocol Violation | 1 | 0
Period: Period 2: 100 mg Vorinostat
Arm/Group | Vorinostat 200 mg | Vorinostat 100 mg
Started | 0 | 6
Completed | 0 | 5
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Arm/Group | Vorinostat, 5-FU, Radiation Therapy
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 2
Age, Continuous [Median (Full Range); unit: years] | 60.7 [48.2 to 78.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Maximally Tolerated Dose (MTD) of Vorinostat in Combination With Infusional 5-FU and Radiation Therapy.
Description: The maximum tolerated dose (MTD) is defined as one dose level below the dose level at which participants experience an unacceptable rate of dose-limiting toxicity.
Time Frame: 6 weeks
Measure: Number; unit: milligrams per day
Arm/Group | Vorinostat, 5-FU, Radiation Therapy
Number analyzed (Participants) | 10
milligrams per day | NA — Criteria for Maximum Tolerated Dose (MTD) were not met before premature closure of the study and therefore a MTD was not determined.

2. Primary Outcome: Progression Free Survival (PFS) at 7 Months From Registration
Description: Progression free survival was defined as the duration of time from registration on study to time of objective disease progression. Death was regarded as a progression event. Progression was defined by the Response Evaluation Criteria in Solid Tumors (RECIST) as at least a 20% increase in the sum of the longest diameter of target lesions, or the appearance of one or more new lesions as seen on radiologic evaluation.
Time Frame: 7 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Vorinostat, 5-FU, Radiation Therapy
Number analyzed (Participants) | 10
months | NA [1.74342 to NA] — The estimated survival probability never reached 50% during 7 months of follow-up, so the median and 95% CI could not be calculated.

3. Secondary Outcome: Progression Free Survival
Description: Progression free survival for this endpoint was defined as the duration of time from beginning of the patients' initial chemotherapy to time of objective disease progression. Death was regarded as a progression event. Progression was defined by the Response Evaluation Criteria in Solid Tumors (RECIST) as at least a 20% increase in the sum of the longest diameter of target lesions, or the appearance of one or more new lesions as seen on radiologic evaluation.
Time Frame: 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Vorinostat, 5-FU, Radiation Therapy
Number analyzed (Participants) | 10
months | 9.375 [1.7434 to 13.7829]

4. Secondary Outcome: Number of Participants Experiencing Unacceptable Toxicity
Description: All participants who receive at least one dose of study treatment were evaluable for toxicity. Unacceptable toxicity is based on the Common Terminology Criteria for Adverse Events (CTCAE) version 3.0. Most grade 3 (severe) or 4 (life-threatening) events are considered to be unacceptable toxicities -- exceptions include nausea or vomiting, fatigue, and alopecia. Hematologic toxicities need to be either grade 4 or last for protocol-defined durations to be considered unacceptable.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Vorinostat 200 mg | Vorinostat 100 mg
Number analyzed (Participants) | 4 | 6
Participants | 1 | 1

5. Secondary Outcome: Overall Survival
Description: Percentage of participants still alive at 1 year after enrollment on study
Time Frame: 1 year
Population: One participant excluded from this analysis due to non-compliance with study drug administration.
Measure: Count of Participants; unit: Participants
Arm/Group | Vorinostat, 5-FU, Radiation Therapy
Number analyzed (Participants) | 9
Participants | 6

6. Secondary Outcome: Response Rate
Description: Participants who have either a complete response (disappearance of all target lesions), partial response (at least 30% decrease in sum of longest diameter of target lesions) or stable disease (decrease in size of less than 30% or increase in size of less than 20%).
Time Frame: 1 year
Population: One participant excluded from this analysis due to non-compliance with study drug administration.
Measure: Count of Participants; unit: Participants
Arm/Group | Vorinostat, 5-FU, Radiation Therapy
Number analyzed (Participants) | 9
Participants | 6

7. Secondary Outcome: Resectability Rate
Description: Percentage of patients able to undergo surgical resection after protocol therapy.
Time Frame: 5 months
Population: One participant excluded from this analysis due to non-compliance with study drug administration.
Measure: Count of Participants; unit: Participants
Arm/Group | Vorinostat, 5-FU, Radiation Therapy
Number analyzed (Participants) | 9
Participants | 2

ADVERSE EVENTS:
Time Frame: Approximately 3 months. Any events experienced while on study medication, throughout the study, and within 30 days of the last dose of study medication.
Description: Information on all adverse events, whether reported by the participant, directly observed, or detected by physical examination, laboratory test or other means, will be collected, recorded, followed and reported.
Groups:
- Vorinostat 200mg: Vorinostat 200 mg; orally, days 1-7, weeks 1-6 5-FU 225 mg/m2/day; intravenous over 24 hours; days 1-5, weeks 1-6 until completion of radiation therapy; Radiation therapy; 180cGy daily Monday-Friday; 28 days of treatment (6 weeks)during each week of radiation therapy
- Vorinostat 100mg: Vorinostat 100 mg; orally, days 1-7, weeks 1-6 5-FU 225 mg/m2/day; intravenous over 24 hours; days 1-5, weeks 1-6 until completion of radiation therapy; Radiation therapy; 180cGy daily Monday-Friday; 28 days of treatment (6 weeks)
Arm/Group | Vorinostat 200mg | Vorinostat 100mg
Serious Adverse Events (participants affected / at risk) | 1/4 | 1/6
Other Adverse Events (participants affected / at risk) | 4/4 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vorinostat 200mg (N=4) | Vorinostat 100mg (N=6)
Disease Progression NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Dehydration (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vorinostat 200mg (N=4) | Vorinostat 100mg (N=6)
Hemoglobin (Investigations) | 1 (1) | 3 (3)
Leukocytes (Investigations) | 3 (3) | 2 (2)
Lymphopenia (Investigations) | 3 (3) | 6 (6)
Neutrophils (Investigations) | 1 (1) | 0 (0)
Platelets (Investigations) | 1 (1) | 4 (4)
Arrhythmia-other (Cardiac disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 4 (4) | 6 (6)
Fever w/o neutropenia (General disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Rigors/chills (General disorders) | 1 (1) | 1 (1)
Weight gain (Investigations) | 0 (0) | 1 (1)
Weight loss (Investigations) | 3 (3) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (2)
Hand-foot reaction (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
Skin-other (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 3 (3) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 2 (2) | 1 (1)
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (4) | 4 (4)
Stenosis (incl anastomotic) biliary tree (Hepatobiliary disorders) | 0 (0) | 1 (1)
Taste disturbance (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nose, hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Infection Gr0-2 neut, upper airway (Infections and infestations) | 1 (1) | 1 (1)
Edema limb (General disorders) | 2 (2) | 0 (0)
Lymphatics-other (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Alkaline phosphatase (Investigations) | 1 (1) | 1 (1)
ALT, SGPT (Investigations) | 0 (0) | 2 (2)
AST, SGOT (Investigations) | 1 (1) | 3 (3)
Bicarbonate (Investigations) | 1 (1) | 1 (1)
Bilirubin (Investigations) | 0 (0) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Creatinine (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 4 (4)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 2 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Neuropathy-sensory (Nervous system disorders) | 0 (0) | 1 (1)
Abdomen, pain (Gastrointestinal disorders) | 0 (0) | 3 (3)
Back, pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Extremity-limb, pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain-other (General disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
Only 10 participants were enrolled on this trial that planned for 50. Phase II portion of the study was not reached and therefore endpoint analysis is severely limited by sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes